CLINICAL TRIAL: NCT01304693
Title: Safety and Efficacy Study of ESBA1008 Versus LUCENTIS® for the Treatment of Exudative Age-Related Macular Degeneration
Brief Title: ESBA1008 Safety, Tolerability and Effects in Wet Age-Related Macular Degeneration (AMD) Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-10-083
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Exudative Age-Related Macular Degeneration
Keywords: AMD; Wet AMD; Exudative; CNV
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ESBA1008 (Experimental): ESBA1008 solution, single intravitreal injection
  Interventions: Biological: ESBA1008 solution
- LUCENTIS (Active Comparator): Ranibizumab 0.5 mg, single intravitreal injection
  Interventions: Biological: Ranibizumab 0.5 mg

INTERVENTIONS:
Biological: ESBA1008 solution — Administered as a single intravitreal injection (Dose A, Dose B, Dose C, Dose D)
  Arms: ESBA1008
Biological: Ranibizumab 0.5 mg — Administered as a single intravitreal injection
  Other Names: LUCENTIS®
  Arms: LUCENTIS

SUMMARY:
The purpose of this study was to assess the safety, tolerability, and the effects of treatment on ocular outcomes following a single intravitreal administration of ESBA1008 compared with LUCENTIS® in patients with exudative age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
This study was conducted in two parts. In Part 1, patients were initially randomized (5:2) to receive either ESBA1008 at the lowest dose (Dose A) or LUCENTIS. After Safety Committee review, a second cohort was enrolled and randomized (5:2) to the next higher dose of ESBA1008 (Dose B). Safety review and enrollment of patients into the third cohort (Dose C) and fourth cohort (Dose D) was conducted in the same manner. Part 2, the expansion period, consisted of 2 arms. In the first arm patients were randomized to receive ESBA1008 Dose C or LUCENTIS (43:44) . In the second arm, patients were randomized to ESBA1008 Doses A:B:D:Lucentis (5:30:35:9). All enrolled patients (Part 1 and Part 2) were evaluated for safety and efficacy across 13 study visits, including Screening, Randomization, and 11 post- treatment follow-up visits (Day 1 through Month 6).

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Primary subfoveal choroidal neovascularization (CNV) secondary to AMD, including predominantly classic, minimally classic or occult lesions, in the study eye.
* New diagnosis of wet AMD or evidence of recent disease progression within the last 3 months in study eye.
* Evidence of subretinal fluid or retinal cystic changes with a CSFT of > 340 μm using a Spectralis SD-OCT (Heidelberg Engineering) imaging system.
* Best-corrected visual acuity (BCVA) of Snellen equivalent 20/200 or better in the non-study eye.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Previously administered therapy, approved or investigational, for wet AMD in the study eye.
* Any current or history of macular or retinal disease in the stuy eye other than wet AMD.
* Lasik or cataract surgery within the last 3 months in the study eye or expected to have cataract removal surgery during the study.
* Uncontrolled or advanced glaucoma in the study eye.
* Use of systemic or topical ocular corticosteroids.
* History of a medical condition that, in the opinion of the Investigator, would preclude scheduled visits, completion of the study, or safe administration of study medication.
* Abnormal or unsuitable laboratory results at Screening visit.
* Lactating or pregnant. Women of childbearing potential must use adequate birth control for the duration of the study.
* Other protocol-defined exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2010-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georges Weissgerber, MD, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 51 investigational centers located in the United States, Europe, Israel, and Australia.
Pre-assignment Details: Of the 376 enrolled, 182 were exited as screen failures prior to exposure to randomization and exposure to the study drug. This reporting group includes all patients who were randomized, received study drug, and completed at least 1 scheduled on-therapy study visit (ITT) (194).
Groups:
- ESBA1008 Dose A; ESBA1008 Dose B; ESBA1008 Dose C; ESBA1008 Dose D; Lucentis: Single intravitreal injection with 6-month follow-up
Period: Overall Study
Arm/Group | ESBA1008 Dose A | ESBA1008 Dose B | ESBA1008 Dose C | ESBA1008 Dose D | Lucentis
Started | 10 | 35 | 48 | 40 | 61
Completed | 10 | 35 | 47 | 39 | 60
Not Completed | 0 | 0 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Decision Unrelated to an Adverse Event | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all patients who were randomized, received study drug, and completed at least 1 scheduled on-therapy study visit (ITT).
Groups:
- Total: Total of all reporting groups
Arm/Group | ESBA1008 Dose A | ESBA1008 Dose B | ESBA1008 Dose C | ESBA1008 Dose D | Lucentis | Total
Number analyzed (Participants) | 10 | 35 | 48 | 40 | 61 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] — This analysis population includes all patients who were randomized, received study drug, and completed at least 1 scheduled on-therapy study visit (Intent-to-Treat).
  years | 75.9 (6.9) | 78.5 (8.3) | 75.2 (7.7) | 74.5 (9.8) | 77.8 (8.1) | 76.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 15 | 27 | 25 | 33 | 106
  Male | 4 | 20 | 21 | 15 | 28 | 88

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Month 1 in Central Subfield Thickness (CSFT) as Measured by Spectral Domain Ocular Coherence Tomography (SD-OCT)
Description: CSFT is a retinal thickness measurement and was measured with SD-OCT. A thickening of the retina is characteristic of wet AMD, and a reduction in CSFT may indicate an improvement in ocular health. One eye (ie, study eye) contributed to the mean.
Time Frame: Baseline, Month 1
Population: This analysis population includes all patients who were randomized, received study drug, and completed at least 1 scheduled on-therapy study visit (ITT). Efficacy data from visits occurring after standard of care (SoC) were censored and replaced based on LOCF,i.e. by the data observed at the time of the SoC decision.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | ESBA1008 Dose A | ESBA1008 Dose B | ESBA1008 Dose C | ESBA1008 Dose D | Lucentis
Number analyzed (Participants) | 10 | 35 | 48 | 40 | 61
microns | -142.3 (78.8) | -181.6 (107.2) | -175.6 (138.9) | -174.9 (101.3) | -159.4 (110.1)

2. Secondary Outcome: Duration of Effect Measured by the Time From Randomization to Receipt of Standard of Care as Determined by the Investigator Based on Protocol Criteria
Description: Standard of care (SOC) therapy for exudative AMD was implemented if any protocol-specified criteria relating to CSFT, best-corrected visual acuity, or clinically significant intraocular hemorrhages in the study eye were met, in the opinion of the Investigator.
Time Frame: Time to event, up to Month 6
Population: ITT: All patients who were randomized, received study drug, and completed at least 1 scheduled on-therapy study visit.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | ESBA1008 Dose A | ESBA1008 Dose B | ESBA1008 Dose C | ESBA1008 Dose D | Lucentis
Number analyzed (Participants) | 10 | 35 | 48 | 40 | 61
Days | 45 [30 to 60] | 75 [45 to 120] | 67.5 [37.5 to 120] | 75 [37.5 to 150] | 45 [25 to 75]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (2 years, 5 months). An AE was considered to be any untoward medical occurrence in a patient exposed to study drug. The AE did not have to have had a causal relationship with the study drug.
Description: This analysis population includes all patients exposed to the study drug, as treated. It should be noted that 6 patients were misdosed: 1 randomized to ESBA1008 B received ESBA1008 A; 1 randomized to ESBA1008 C received ESBA1008 B; and 4 randomized to ESBA1008 B received ESBA1008 D.
Arm/Group | ESBA1008 Dose A | ESBA1008 Dose B | ESBA1008 Dose C | ESBA1008 Dose D | Lucentis
Serious Adverse Events (participants affected / at risk) | 0/11 | 4/31 | 3/47 | 3/44 | 7/61
Other Adverse Events (participants affected / at risk) | 1/11 | 10/31 | 17/47 | 16/44 | 13/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ESBA1008 Dose A (N=11) | ESBA1008 Dose B (N=31) | ESBA1008 Dose C (N=47) | ESBA1008 Dose D (N=44) | Lucentis (N=61)
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Post-procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Aortic bypass (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Endophthalmitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ESBA1008 Dose A (N=11) | ESBA1008 Dose B (N=31) | ESBA1008 Dose C (N=47) | ESBA1008 Dose D (N=44) | Lucentis (N=61)
Conjunctival haemorrhage (Eye disorders) | 0 | 3 | 3 | 8 | 2
Nasopharnygitis (Infections and infestations) | 1 | 0 | 3 | 3 | 2
Retinal haemorrhage (Eye disorders) | 0 | 1 | 2 | 1 | 4
Visual acuity reduced (Eye disorders) | 0 | 2 | 1 | 2 | 3
Hypertension (Vascular disorders) | 0 | 1 | 5 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 4 | 1 | 2 | 0
Eye pain (Eye disorders) | 0 | 0 | 4 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 3 | 0 | 3
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.